CLINICAL TRIAL: NCT03454347
Title: The Efficacy of Protein Supplementation on Attenuating Muscle Atrophy Following Disuse in the Collegiate Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Dakota State University (Other)
Collaborators: Sanford Research (Other)
Responsible Party: Principal Investigator, Lee Weidauer, Assistant Professor, South Dakota State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-1801014-EXP
Record Dates: First submitted 2018-02-22; First posted 2018-03-05 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Disuse Atrophy
MeSH Terms: conditions — Muscular Disorders, Atrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein Supplementation Group (Experimental): Participants in this group will complete two weeks of lower limb suspension and receive 75g/day of supplemental protein in addition to education aimed at increasing protein intake through their diet.
  Interventions: Dietary Supplement: Profile Perform
- Non-Supplemental Group (Active Comparator): Participants in this group will complete two weeks of lower limb suspension and will receive no supplementation or nutritional education.
  Interventions: Other: Lower Limb Suspension

INTERVENTIONS:
Dietary Supplement: Profile Perform — The dietary supplement includes 1.5 grams of fat, 19 grams of carbohydrate, and 25 grams of protein per serving. Participants in the experimental group will consume 3 servings per day.
  Arms: Protein Supplementation Group
Other: Lower Limb Suspension — This group will complete two weeks of lower limb suspension.
  Arms: Non-Supplemental Group

SUMMARY:
Following orthopedic surgery and/or injury, a significant loss of muscle mass is generally observed. While this loss of muscle mass appears to be the norm, it causes significant problems in both the athletic and general population. Athletes struggle to regain their performance because of the decrease in muscle mass and also have a greater potential for reinjury while they are in a depleted state. In the general population, and particularly among the elderly, this loss in muscle mass can be even more devastating because as people age, it is more difficult to regain muscle after it is lost. In elderly individuals, this loss in muscle mass can lead to significant disability, diminished quality of life along with an increased risk of falls. In addition to the muscle mass lost during the post-operative period, the strength of the muscle also decreases. This has obvious performance implications in athletes, as well as having the potential to extend recovery time. In the elderly, decreased strength may result in reduced independence and inability to perform activities of daily living. Many previous bed rest studies have reported that significant bone loss also occurs during times of decreased mechanical loading. The post-operative period generally results in decreased mechanical loading; however, some muscle loading will still occur during the rehabilitation process. The dynamic relation between muscle activity/loading and bone density changes in the post-operative state has not been fully described and requires further study.

With this knowledge of the importance of nutrition to the musculoskeletal system, applying the principles of increased protein intake through the addition of a dietary supplement to a population preparing for orthopedic surgery and subsequent muscle disuse is a logical next step. The investigators hypothesize that through the consumption of a protein-based dietary supplement three times per day (75g protein), along with educating patients on the importance of consuming foods that are high in protein, there will be an attenuation of decreases in muscle mass and strength as well as losses in bone that occur with orthopedic injury and disuse. The investigators long-term goal is to identify a nutritional protocol that can be implemented prior to and following orthopedic surgery to diminish the deleterious effects of the subsequent disuse on muscle and bone.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be physically active males and females aged 18-25 with no history of a lower extremity injury 12 months prior to participation. Physically active will be classified as participating in physical activity for at least 3 minutes and a minimum of 3 days per week.

Exclusion Criteria:

* Participants will be excluded if they are participating in any other research projects that could potentially affect the outcomes of this study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Muscle Mass | Measurements will be obtained prior to immediately following 2 weeks of lower limb suspension
  Whole body muscle mass (kg) will be measured using DXA while muscle cross-sectional area of the lower leg will be measured via pQCT

SECONDARY OUTCOMES:
Muscle strength | Measurements will be obtained prior to immediately following 2 weeks of lower limb suspension
  Torque production (NM) will be measured using isokinetic testing with a Biodex System 4 Ergometer. The protocol will include maximal quadricep extension and hamstring flexion performed at 60, 180, and 300 degrees per second

OTHER OUTCOMES:
Volumetric bone mineral density | Measurements will be obtained prior to immediately following 2 weeks of lower limb suspension
  Volumetric bone mineral density (mg/cm^2) at the 66% slice of the tibia will be measured using pQCT
Bone Cross-Sectional Area | Measurements will be obtained prior to immediately following 2 weeks of lower limb suspension
  Total bone cross sectional area (cm^2) at the 66% slice of the tibia will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- South Dakota State University, Brookings, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No